CLINICAL TRIAL: NCT03193333
Title: A Non-inferiority in the Intraocular Pressure Decrease of the Preservative-free Ophthalmic Solution PRO-122 Versus Concomitant Therapy in Subjects With Uncontrolled Primary Open-angle Glaucoma
Brief Title: PRO-122 Versus Concomitant Therapy in Subjects With Uncontrolled Primary Open-angle Glaucoma (PRO-122LATAM)
Acronym: PRO-122LATAM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's prerogative since initial purpose for study shifted according to business strategy.
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH122-0316/III
Record Dates: First submitted 2017-06-19; First posted 2017-06-20 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Primary Open-angle Glaucoma
Keywords: glaucoma; primary open-angle glaucoma; Ophthalmic antihypertensives; Krytantek Ofteno®.; timolol; brimonidine; dorzolamide
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Timolol; Brimonidine Tartrate; dorzolamide

STUDY DESIGN:
Intervention Model Description: A non-inferiority, phase III, double-blind, randomized, controlled, parallel, clinical trial
Who Masked: Participant, Investigator
Masking Description: Blinding will be performed by the personnel assigned by the Laboratorios Sophia S.A. de C.V. Clinical Operations Management. The blinding will consist in the elimination of the primary label (commercial) for Krytantek Ofteno® and the triple concomitant therapy and the placement of a label identical to those of the other interventions. Since the bottles in which Krytantek Ofteno® and the concomitant therapies are different in color and cap shape to the ones used for the placebo and the PRO-122, a masking will be performed in the primary packaging, which shall be identical for all three interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRO-122 group (Experimental): To validate the 3 flasks of the triple therapy will be used 1 bottle with the three active principles (PRO-122) and two placebos and thus comply with the masking.
  Drug substances: Timolol 5 mg/mL, brimonidine 2 mg/mL and dorzolamide 20 mg/mL. preservative free.
  Pharmaceutical form: Ophthalmic solution
  Made by: Laboratorios Sophia, S.A. de C.V.
  Posology: 1 drop every 12 hours for 90 days
  Description of the solution: clear, visibly particle free, slightly yellow solution, preservative free
  * Package description: 5 m multidose dropper bottle.
    * Placebo (for
  * Two pieces of approved placebo. Administered in 2 multidose dropper bottles.
  * Posology: 1 drop of each dropper bottle every 12 hours for 90 days
  Interventions: Drug: PRO-122; Other: Placebo1; Other: Placebo 2
- Concomitant triple therapy group (Active Comparator): Imot Ofteno
  Drug substance: Timolol 5 mg/mL
  Pharmaceutical form: Ophthalmic solution
  Made by Laboratorios Sophia S.A. de C.V.
  Alphagan
  Drug substance Brimonidine 2 mg/mL
  Pharmaceutical form: Ophthalmic solution
  Made by: Allergan, Inc.
  Trusopt
  Drug substance: Dorzolamide 20 mg/mL
  Pharmaceutical form: Ophthalmic solution
  Made by: Merck Sharp and Dohme Corp.
  Posology: 1 drop every 12 hours for 90 days
  Interventions: Drug: Timolol eye drops; Drug: Dorzolamide-Timolol Ophthalmic; Drug: Brimonidine Ophthalmic Solution
- Krytantek Ofteno Group (Active Comparator): To validate the three flasks of the triple therapy will be used 1 bottle with the three active principles (Krytantek) and two placebos and thus comply with the masking.
  Drug substances: Timolol 5 mg/mL, brimonidine 2 mg/mL and dorzolamide 20 mg/mL.
  Pharmaceutical form: Ophthalmic solution
  Made by: Laboratorios Sophia, S.A. de C.V.
  Posology: 1 drop every 12 hours for 90 days
  Description of the solution: clear, visibly particle free, slightly yellow solution Package description: 5 m multidose dropper bottle.
  Placebo (for two pieces of approved placebo. Administered in 2 multidose dropper bottles.
  Posology: 1 drop of each dropper bottle every 12 hours for 90 days
  Interventions: Other: Placebo1; Other: Placebo 2; Drug: Krytantek

INTERVENTIONS:
Drug: PRO-122 — Posology: 1 drop every 12 hours for 90 days
  Other Names: krytantek PF (Timolol, Brimonidine, Dorzolamide)
  Arms: PRO-122 group
Drug: Timolol eye drops — 1 drop every 12 hours for 90 days
  Other Names: Concomitant triple therapy
  Arms: Concomitant triple therapy group
Drug: Dorzolamide-Timolol Ophthalmic — 1 drop every 12 hours for 90 days
  Other Names: Concomitant triple therapy
  Arms: Concomitant triple therapy group
Drug: Brimonidine Ophthalmic Solution — 1 drop every 12 hours for 90 days
  Other Names: Concomitant triple therapy
  Arms: Concomitant triple therapy group
Other: Placebo1 — 1 drop of each dropper bottle every 12 hours for 90 days
  Arms: Krytantek Ofteno Group; PRO-122 group
Other: Placebo 2 — 1 drop of each dropper bottle every 12 hours for 90 days
  Arms: Krytantek Ofteno Group; PRO-122 group
Drug: Krytantek — Posology: 1 drop every 12 hours for 90 days
  Arms: Krytantek Ofteno Group

SUMMARY:
Objectives: To evaluate the non-inferiority in the intraocular pressure decrease of the preservative-free ophthalmic solution PRO-122, manufactured by Laboratorios Sophia S.A. de C.V., versus concomitant therapy in subjects with uncontrolled primary open-angle glaucoma and/or IOP.

Hypothesis: The mean (average) value of the IOP final absolute reduction in the experimental group (PRO-122) is not lower, considering a lower limit of 1 mmHg, compared to the IOP mean absolute reduction of the standard group (concomitant therapy).

Methodology: A non-inferiority, phase III, double-blind, randomized, controlled, parallel, clinical trial

DETAILED DESCRIPTION:
Number of patients: 51 subjects divided into 3 groups (17 subjects per group)

Diagnosis and main inclusion criterion:

Diagnosis: Primary open-angle glaucoma or ocular hypertension

Main criteria:

* Patients of either sex
* Average intraocular pressure (IOP) ≤ 36 mm/Hg
* Previous management with ocular hypotensive medications ≥ 2 months, without achieving control (target IOP)
* Age ≥ 18 years
* Informed consent

Test product, dosage and route of administration:

* PRO-122. Preservative-free ophthalmic solution of timolol 0.5% / brimonidine 0.2% / dorzolamide 2% Manufactured by Laboratorios Sophia, S.A. de C.V., Zapopan, Jalisco, Mexico. + Placebo + Placebo
* Dosage: 1 drop every 12 hours
* Route of administration: ophthalmic

Treatment duration: 90 days

Evaluation criteria:

Efficiency (non-inferiority):

* IOP decrease

Safety:

* Best corrected visual acuity
* Cup-to-disc ratio
* Visual fields determined by computerized perimetry
* Central corneal thickness determined by pachymetry
* Ocular surface integrity, including:

  * Conjunctival hyperemia
  * Chemosis
  * Fluorescein staining
* Density of goblet cells
* Adverse events

Tolerability:

* Ocular comfort index

Statistical methodology:

The data will be expressed with measures of central tendency: mean and standard deviation for quantitative variables. The qualitative variables will be presented in frequencies and percentages. Statistical analysis will be done by means of a Kruskal-Wallis test for quantitative variables. The difference between qualitative variables will be analyzed using an square chi An alpha ≤ 0.05 would be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age greater or equal to 18 years
* Both sexes
* Women of childbearing age with birth control method
* Diagnosis of Primary open-angle glaucoma (according to the Guidelines of the Preferred Practice Pattern of the American Academy of Ophthalmology) or ocular hypertension (OHT)
* Intraocular pressure (IOP) not controlled with dual therapy according to the principal investigator (PI) judgment.
* IOP on the selection visit at 9 am, after the washing period, from 21 - 36 mmHg in at least one eye.

Exclusion Criteria:

General criteria

* Pregnant, breastfeeding or planning to get pregnant women.
* Women of childbearing age and who do not intake a hormonal contraceptive method, intrauterine device or bilateral tubal obstruction.
* Participation in another clinical research study greater or equal 30 days before the screening visit.
* People who cannot comply with their attendance at appointments or with all the - Protocol requirements

Medical and therapeutic criteria:

* Anterior chamber angle grade less than 2 of Shaffer rating.
* Excavation of optic nerve greater than 0.80 horizontal or vertical (ratio cup-disc)
* Serious loss of central visual field in any eye (sensitivity less or equal to 10 decibels in greater or equal to 2 of 4 points of the visual field test close to the fixation point)
* People not able to safely suspend ocular hypotensives drug products for the washout period according to the PI judgement.
* Chronic, recurrent, or active ocular inflammatory diseases (e.g. uveitis, scleritis, keratitis, herpetic) in any eye.
* Eye trauma less or equal to 6 months prior to the study
* Eye infection / inflammation less or equal to 3 months prior to the study
* Clinically significant or progressive retinal disease (e.g. degenerations, diabetic retinopathy, retinal detachment)
* Ability Visual 20/200 or worse in any of the eyes.
* Subject with only one eye
* Eye diseases that contraindicate the use of Beta-blocker (BB) Alpha-adrenergic agonist (AA) or Carbonic anhydrase inhibitors (CAIs)
* Intraocular surgery less or equal to 6 months prior to the study
* Laser intraocular surgery less or equal to 3 months prior to the study
* Any abnormality preventing reliable applanation tonometry
* Unstable or uncontrolled cardiovascular disease
* Chronic pulmonary disease (e.g. bronchial asthma)
* Any condition or illness that do not fit the subject for the study according to the PI judgment.
* Use of high doses of salicylate (1 g daily) less or equal to4 weeks before the eligibility visit
* In treatment with psychotropic medications that increase the adrenergic response
* Known hypersensitivity to BB medications (e.g. timolol), AA (e.g. brimonidine) and CAI (e.g. dorzolamide), sulfonamide derivatives, or any of the components of the study drugs
* Concomitant use of monoamine oxidase inhibitors
* Systemic or topical use of corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
intraocular pressure (IOP) | 90days
  Intraocular pressure, Unit: Millimeters of mercury (mmHg) type of variable: Continuous, Measurement method: Goldman applanation tonometry. Normal intraocular pressure 11-21 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (2):
- MD. Sandra Belalcazar Rey, Bogotá, Bogota D.C., Colombia
- MD. Victoria Eugenia Sanchez Castellanos, Zapopan, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT03193333/Prot_SAP_001.pdf